CLINICAL TRIAL: NCT06168643
Title: Effects of Core Stability Exercises With And Without Pregnancy Support Belt On Pain, Function And Disability In Symphysis Pubis Dysfunction During Pregnancy.
Brief Title: Effects of Core Stability Exercise With Pregnancy Support Belt in Pubic Symphysis Dysfunction.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Principal Investigator, Adeela Arif, Senior Lecturer, Riphah International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ayesha Sarwar
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Symphysis Pubis Dysfunction
Keywords: Pain; pregnancy; Exercise; Symphysis pubis dysfunction
MeSH Terms: conditions — Pelvic Girdle Pain; Pain; Motor Activity | interventions — Core Stability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core stability (Experimental)
  Interventions: Other: Core stability
- Core stability with pregnancy support belt (Experimental)
  Interventions: Other: Core stability with pregnancy support belt

INTERVENTIONS:
Other: Core stability — Physical therapy interventions will include core stability exercises which will be demonstrated and will be checked if they are being performed correctly. The exercises guided shall be performed 3 times daily and logbook will be provided to keep the record of exercise program.
  Arms: Core stability
Other: Core stability with pregnancy support belt — Participants will receive same information and exercises as those in Group A. they will also receive pregnancy support belt. The logbook will be provided to keep the record of hours the belt has been worn along with exercise record.
  Arms: Core stability with pregnancy support belt

SUMMARY:
Symphysis pubic dysfunction is a well-known clinical problem encountered by many females during pregnancy, yet it has not received much attention in the research literature. As pubic symphysis dysfunction at times presents with severe pain while performing day to day activities and also affects significantly on quality of life in antenatal period, but its effective management remains difficult to determine as no standardized treatment protocols are available. This study may add to the growing body of knowledge in the management of SPD, that if the core stability exercise alone or with the pregnancy support belts yield comparable outcomes and if one technique is superior to the other, which should be the alternative choice of therapy.

DETAILED DESCRIPTION:
The study will be a randomized clinical trial and will be conducted in Women Care Clinic, Bahawalpur. This study will be completed in time duration of 10 months after the approval of synopsis. Non-probability convenience sampling technique will be used and participants will be recruited in study after randomization. The subjects will be divided into two groups. Group A will receive core stability exercises and group B will receive core stability exercises along with pregnancy support belt. The data will be assessed at the baseline and after 6th week of treatment. After data collection, the data will be analyzed by using SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

Age 25-35 years females Have pain in the region of pubic symphysis, with or without radiation to the groin.

Have pain during stair climbing, turning over in bed, standing on one leg. Have tenderness on palpation of symphysis pubis. Have positive active straight leg raise (ASLR) test result

Exclusion Criteria:

Medical conditions preventing use of pregnancy support belts. Pregnant females having SPD but with absolute contraindications to exercise. Posterior (lumber spine or sacroiliac joint) pain that was considered worse than the symphysis pubis pain

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Roland-Morris Questionnaire (modified) | 6th week
  Roland-Morris Disability Questionnaire (RMDQ) is designed to assess self-rated physical disability caused by low back pain. This scale is used on subjects of age more than 12 years. Each question is worth one point so score can range from 0 (no disability) to 24 (severe disability).
Numerical pain rating scale | 6th week
  The Numerical pain rating scale is the most commonly used pain scale in the health care. This scale is used on subjects of age more than 9. By using this scale ask the participant to rate their pain orally by giving the numbers from 0-10
Pain Specific Functional Scale | 6th Week
  The PSFS is a self-reported valid, reliable, and responsive outcome measure for patients with musculoskeletal problems. Patients are asked to identify up to five important activities they are unable to perform and rate (on an 11-point scale) the current level of difficulty associated with each activity."0" represents "unable to perform" and "10" represents "able to perform at prior level

CONTACTS AND LOCATIONS:
Locations (1):
- Riphah International university, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jain S, Eedarapalli P, Jamjute P, Sawdy R. Symphysis pubis dysfunction: a practical approach to management. The Obstetrician & Gynaecologist. 2006;8(3):153-8.
- [Background] Depledge J, McNair PJ, Keal-Smith C, Williams M. Management of symphysis pubis dysfunction during pregnancy using exercise and pelvic support belts. Phys Ther. 2005 Dec;85(12):1290-300. PMID 16305268
- [Background] MacLennan AH, MacLennan SC. Symptom-giving pelvic girdle relaxation of pregnancy, postnatal pelvic joint syndrome and developmental dysplasia of the hip. The Norwegian Association for Women with Pelvic Girdle Relaxation (Landforeningen for Kvinner Med Bekkenlosningsplager). Acta Obstet Gynecol Scand. 1997 Sep;76(8):760-4. doi: 10.3109/00016349709024343. PMID 9348254